CLINICAL TRIAL: NCT04261946
Title: Post Operative Quality of Life Assesment After Patulous Eustachian Tube Surgical Treatment
Brief Title: Post Operative Quality of Life After Patulous Eustachian Tube Treatment
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-PT-01
Record Dates: First submitted 2019-11-20; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-11

CONDITIONS: Eustachian Tube Patulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life survey — Unilateral patulous eustachian tube surgically treated were interviewed about our life's quality by a survey

SUMMARY:
Patulous eustachian tube (ET) is a usually asymptomatic poorly known ET pathology. When it becomes so and thus impairs the eardrum (retraction pockets, cholesteatoma) or patients' quality of life (QoL), therapeutic management is proposed. The surgical treatment has diversified in recent years but remains dominated by filling spaces around the ET (autologous fat and/or septal cartilage grafting). Efficiency is traditionally objectivized by dynamic otoscopy, tubomanometry and audiometry, but QoL must also be taken into account and its postoperative assesment was the objective of this work.

Materials and Methods This is a unicentric retrospective study conducted from November 2016 to March 2019 on all patients with a disabling patulous ET, single or bilateral, managed surgically by autologous fat and/or septal cartilage grafting in investigators ENT department. Patients for whom a concomitant procedure was performed were excluded from the study.

The post-operative QoL assessment was performed using the Glasgow Benefit Inventory (GBI), postoperative self-administered questionnaire validated in ENT, including a general, physical and social evaluation. Predictive factors for QoL improvement were investigated among pre-, per- and post-operative clinical data.

ELIGIBILITY:
Inclusion Criteria:

* any surgically treateble patient with a unilateral patuluos eustachian tube

Exclusion Criteria:

* any patient for whom an other surgical step than the eustachian tube one was needed,
* bilateral desease ,cholesteatoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient consulting in IUFC (NICE) with a unilateral disabling patulous eustachian tube surgically treated
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Postoperative quality of life | quality of life score in beetwen 2 and 12 month postoperatively
  glasgow benefit inventory : Post-operative quality of life score concerning general, social, and physical aspects " studied in 18 questions. A likert scale ranging from -2 to +2 (5 points) evaluate each of 18 points. Positive and higher score mean a better outcome (maximum = 36). Negative and lower score mean a wors outcome (minimum = -36).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de la Face et du Cou, Nice, France

IPD SHARING:
Plan to Share IPD: No